CLINICAL TRIAL: NCT02162290
Title: Comparison Between Moderate-high Interval Exercise and Moderate Continuous Exercise in an Advanced Cardiac Rehabilitation Program - Nine Months Follow up
Brief Title: Comparison Between Moderate-high Interval Exercise and Moderate Continuous Exercise in an Advanced Cardiac Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2*175/10
Record Dates: First submitted 2014-06-11; First posted 2014-06-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval exercise (Experimental): Exercise bouts in low and high intensities
  Interventions: Other: Interval exercise training
- Continuous exercise (Experimental): Exercise continuously with moderate intensity
  Interventions: Other: Continuous exercise training

INTERVENTIONS:
Other: Interval exercise training — Exercise bouts in low and high intensities
  Arms: Interval exercise
Other: Continuous exercise training
  Arms: Continuous exercise

SUMMARY:
The research will study the differences between interval training and continuous training among cardiac patients in a cardiac rehabilitation facility.

The main objectives are:

1. Functional capacity measures (VO2 max).
2. Cardiac risk factors
3. Quality of life assessments.

Study hypothesis:

Interval training will be more effective in improving functional capacity, cardiac risk factors and quality of life, compared to continuous training.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone:

  * Myocardial infarction
  * Percutaneous transluminal coronary angioplasty
  * Coronary artery bypass graft

Exclusion Criteria:

* Patients with:

  * Severe ischemia or angina
  * Implantable cardioverter-defibrillator
  * Pacemakers transplants
  * Severe left ventricular dysfunctions
  * Uncontrolled arrhythmias

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximal functional capacity | 9 months
  Outcome is assessed at baseline, after 3 months and at nine months

CONTACTS AND LOCATIONS:
Overall Officials: Yael Pernick, Principal Investigator — Asaf Harofe Medical Center; Zyssman, MD, Study Director — Asaf Harofe Medical Center; Jonathan Moore, PhD, Study Director — Bangor University; Zvi Vered, MD, Study Director — Asaf Harofe Medical Center
Locations (1):
- Asaf Harofe Medical Center, Beer Yaacov, Israel